CLINICAL TRIAL: NCT06870929
Title: Effect of Different Intraoral Scanning Approaches on the Passive Fit of Mandibular All-on-Four Screw-Retained Frameworks
Brief Title: Accuracy of Full Arch Intraoral Scanning
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Ibrahim Soliman, lecturer at faculty of dentistry Ain-Shams University, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RecIR022544
Record Dates: First submitted 2025-03-03; First posted 2025-03-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Completely Edentulous
Keywords: intraoral scanner; photogrammetry; full arch implant restorations; passive fit; one-screw test; screw resistance test

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Simple splinting-assisted intraoral scanning (Active Comparator): The Medit i600 direct intraoral classical scans will be obtained while applying only a basic simple splinting
  Interventions: Device: The Photogrammetry-assisted intraoral scanning; Device: The modified approach of splinting-assisted intraoral scanning
- modified splinting-assisted intraoral scanning technique (Experimental): The Medit i600 direct intraoral scans will be obtained while applying basic simple splinting along with incorporating a unique tip in the scanning protocol and scanner software
  Interventions: Device: Simple splinting-assisted intraoral scanning
- Photogrammetry-assisted intraoral scanning (Experimental): The Medit i600 will be used to obtain direct intraoral scans while the scan bodies are combined with extra photogrammetry system scanning assistance.
  Interventions: Device: Simple splinting-assisted intraoral scanning

INTERVENTIONS:
Device: The Photogrammetry-assisted intraoral scanning — The Photogrammetry-assisted intraoral scanning; will be executed using the MUA-compatible ioConnect ® photogrammetry system components exactly in the same sequence as recommended by the manufacturer
  Arms: Simple splinting-assisted intraoral scanning
Device: The modified approach of splinting-assisted intraoral scanning — The scan bodies will be mounted over the MUA and loosely connected with a power chain before the Medit scanner single-shot scanning procedure. Using the additional scan option in the Medit scanner software, another single-shot scan will be obtained and superimposed to the first scan yielding a color map that reflects the accuracy of the obtained scan and directs a highly precise final scan.
  Arms: Simple splinting-assisted intraoral scanning
Device: Simple splinting-assisted intraoral scanning — The Medit i600 direct intraoral classical scans will be obtained while applying only a basic simple splinting
  Arms: Photogrammetry-assisted intraoral scanning; modified splinting-assisted intraoral scanning technique

SUMMARY:
Although an intraoral scanner IOS can offer the clinician a completely digital workflow, achieving trustworthy digital scans in edentulous jaws is challenging because of the lack of fixed anatomical landmarks. From this perspective, several methods have been proposed to improve the accuracy of digital scanning, however, related results remain inconclusive, and previously proposed devices have had limitations, such as bulkiness, excessive manufacturing requirements, and poor commercial applicability.

Thus, this study aims to clinically compare the effect of conventional versus photogrammetry intraoral scanning methods on the passive fit of mandibular all-on four screw-retained frameworks.

DETAILED DESCRIPTION:
The current study will be designed to be a crossover, double-blinded randomized clinical trial. Eighteen edentulous patients will be selected to share in the study to be rehabilitated by screw-retained prostheses following the all-on-4 protocol. After guided implant surgery, patients will be immediately restored by screw-retained acrylic provisionals following the traditional denture conversion technique. The definitive prosthesis will be fabricated after osseointegration starting with the intraoral scanning procedure; each patient will be subjected to three different scanning methods that can enhance the existing IOS workflow; for group I, the Medit i600 will be used to obtain direct intraoral scans while the scan bodies are combined with extra photogrammetry system scanning assistance, for group II, Medit i600 direct intraoral scans will be obtained while applying basic simple splinting along with incorporating a unique tip in the scanning protocol and scanner software, for group III, Medit i600 direct intraoral classical scans will be obtained while applying only a basic simple splinting. The STL file obtained from the different scans will be sent directly to the dental laboratory and three CAD/Milled frameworks will be realized based on the acquired scans. The jigs' passivity will be tested in the patient's mouth by the single screw test followed by the screw resistance test and the screw resistance test parameter will be calculated. The results will be collected for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a completely edentulous lower arch that could be restored by fixed screw-retained implant prosthesis.
* Patients having a substantial bone height and width at prospective implant sites to install four standard-size implants following the all-on-4 protocol.
* Patients having Sufficient crown height space.

Exclusion Criteria:

* Patients with bad oral hygiene.
* Patients with limited mouth opening.
* Vulnerable groups.
* Uncooperative patients.
* Patients receiving or undergoing radiotherapy or chemotherapy. Patients with systemic diseases affecting bone metabolism. Smokers.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of passive fit following the latest update of the one screw test | six months
  Three CAD/Milled frameworks for each subject will be realized based on the acquired scans. The passive fit of each framework will be assessed intraorally following the Sheffield test: The test Part I involves checking the fit of the framework using finger pressure then tightening one of the most distal abutment screws. when an accurate horizontal and perpendicular fit viewed under magnification (will be categorized as 3 or excellent). If a slight "shadow" or suspicion of a vertical discrepancy, exists between the framework and abutment, a satisfactory passive fit will be confirmed by part 2 of test; If a suspected fit discrepancy can be closed using a 13mm wide modelling wax strip, representing 20 KN/m2 pressure load without distorting, then the fit is deemed to be clinically acceptable (categorized as 2 or good). If the wax does distort or is unable to close the discrepancy, will be (categorized as 1 or poor). this categorization arbitrarily defined by authors.

SECONDARY OUTCOMES:
objective assessment of clinical passive fit using the screw resistance test parameter | six months
  The screw resistance test will be used to objectively evaluate and compare the passive fit of the three frameworks for each subject by calculating the SR parameter as the difference of the rotation angles of each screw in the passive and the non-passive situations by the formula: SR = SR passive - SR non-passive.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Ain-Shams university, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still study not completed